CLINICAL TRIAL: NCT02545920
Title: Pilot Study to Assess the Effects of Haemodialysis Treatments on Blood Flow to the Ear
Brief Title: To Assess Ear Blood Flow During Dialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0310
Record Dates: First submitted 2015-07-07; First posted 2015-09-10 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Kidney Failure
Keywords: haemodialysis; hypotension
MeSH Terms: conditions — Renal Insufficiency; Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — observational study

SUMMARY:
This is a prospective observational pilot study of patients under the care of the Royal Free Hospital with chronic kidney disease who have been established on regular thrice weekly haemodialysis treatments in a dialysis centre,to measure the changes in blood flow in the ear during haemodialysis.

DETAILED DESCRIPTION:
10 patients, attending for thrice weekly outpatient haemodiafiltration shall be studied during a dialysis session using a CE marked commercially available digital otoscope capable of recording digital videos of the tympanic membrane and ear canal.

Patients will receive standard clinical care and monitoring of their dialysis session, which includes recording of blood pressure and changes in haematocrit and volume status during dialysis and noting patient symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years and older up to 80 years
* Under the care of the Royal Free Hospital with chronic kidney disease and established on regular thrice weekly haemodiafiltration.
* Able to provide written informed consent obtained

Exclusion Criteria:

* Patients unable to provide written informed consent
* Patients using hearing aids
* Patients who have had previous middle ear surgery
* Patients not fulfilling inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic kidney failure attending for regular dialysis treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
change in ear blood flow | day 1 dialysis session
  percentage change in ear blood flow compared to initial ear blood flow

SECONDARY OUTCOMES:
change in blood pressure | day 1 dialysis session
  change in blood pressure in mmHg compared to starting blood pressure
change in haematocrit volume status | day 1 dialysis session
  percentage change in haematocrit
record of hypotensive episodes during dialysis | day 1 dialysis session
  record of nursing interventions including reduction in ultrafiltration volume, administration of intravenous fluids. Use of distress thermometer visual analogue scale to record patient symptoms

CONTACTS AND LOCATIONS:
Overall Officials: andrew davenport, Principal Investigator — UCL Centre for Nephrology, Royal Free Hospital
Locations (1):
- Royal Free Hospital, London, United Kingdom